CLINICAL TRIAL: NCT05093725
Title: CD49 in Optimization The Cologenicity of Mesenchymal Stem Cell Culture Passage
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, samia samir shawky, resident doctor at clinical pathology in Sohag oncology center, Sohag University
Other Study IDs: Soh-med-21-10-01
Record Dates: First submitted 2021-10-13; First posted 2021-10-26 (Actual); Last update posted 2021-10-26 (Actual); Status verified 2021-10

CONDITIONS: Umbilical Cord of Normal Labor

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: flow cytomery — take sample of Wharton jelly and culturing it to know the best time for mesenchymal stem cell growth

SUMMARY:
Human mesenchymal stem cells (MSCs) due to their regenerative and immunomodulatory properties are widely used for the treatment of bone and cartilage damage, cardiovascular, gastrointestinal, autoimmune, neurodegenerative diseases and cancer .It is shown that the use of MSCs in therapy is safe and can be effective .In 2006, the International Society for Cellular Therapy (ISCT) proposed the minimal criteria to define human MSCs. First, MSCs must be plastic-adherent when maintained in the standard culture conditions. Second MSCs must express CD105, CD73 and CD90, and lack expression of CD45, CD34, CD14 or CD11b, CD79a or CD19 and HLA-DR surface molecules.

ELIGIBILITY:
Inclusion Criteria:

normal babies delivered by normal labor

Exclusion Criteria:

diseased or congenital anomalies

Min Age: 1 Day | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: taking umbilical cord of normally labored babies
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2021-11 (Estimated); Primary Completion 2022-06 (Estimated); Study Completion 2022-06 (Estimated)

PRIMARY OUTCOMES:
evaluation the best passage of MSC culture by CD49 surface marker | 7 months
  evaluation the best passage of MSC culture by CD49 surface marker

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag University Hospital, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Lv FJ, Tuan RS, Cheung KM, Leung VY. Concise review: the surface markers and identity of human mesenchymal stem cells. Stem Cells. 2014 Jun;32(6):1408-19. doi: 10.1002/stem.1681. PMID 24578244
- [Background] Madrigal M, Rao KS, Riordan NH. A review of therapeutic effects of mesenchymal stem cell secretions and induction of secretory modification by different culture methods. J Transl Med. 2014 Oct 11;12:260. doi: 10.1186/s12967-014-0260-8. PMID 25304688